CLINICAL TRIAL: NCT03781505
Title: Effect of Intravenous Paracetamol Combination With Caudal Ropivacaine on Quality of Postoperative Recovery in Pediatric Patients Undergoing Hypospadias Repair.A Randomized Controlled Trial.
Brief Title: Intravenous Paracetamol in Combination With Caudal Ropivacaine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Dr. Muhammad Saad Yousuf, Principal Investigator, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 5445-Ane-ERC-18
Record Dates: First submitted 2018-11-23; First posted 2018-12-20 (Actual); Results first posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Analgesia

STUDY DESIGN:
Intervention Model Description: Randomized control trail
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous paracetamol with Caudal Ropivacaine (Experimental): Paracetamol is widely accepted and most commonly used as an adjuvant for postoperative analgesia. It also improves the quality of recovery by attenuating the pain associated with the surgical position. Adverse effects associated with the paracetamol are rare <1/10000, which includes malaise, increased level of hepatic transaminases and hypersensitivity reaction. It has been studied in combination with caudal analgesia with bupivacaine through the rectal route 7,8 with variable results.
  Caudal anaesthesia is effective in alleviating pain below the umbilicus. Also if the caudal block is administered at the beginning of surgery, the effect will start wearing off 2 to 3 hours post surgery. Administration of paracetamol towards end of surgery may help with both these issues. In this study we aim to investigate the effect of adding intravenous paracetamol in combination with caudal analgesia with ropivacaine, hoping that it may improve quality of postoperative analgesia and recovery.
  Interventions: Drug: Paracetamol +caudal ropivacaine
- Placebo (Placebo Comparator): Intravenous Normal Saline with Caudal Ropivacaine
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol +caudal ropivacaine — Paracetamol + Ropivacaine
  Arms: Intravenous paracetamol with Caudal Ropivacaine
Drug: Placebo — Caudal ropivacaine
  Arms: Placebo

SUMMARY:
To investigate whether the addition of intravenous paracetamol with caudal ropivacaine leads to better quality of postoperative recovery in patients undergoing hypospadius repair than caudal ropivacaine alone. The quality of recovery will be judged by postoperative analgesia requirement and lesser agitation in the postoperative period.

DETAILED DESCRIPTION:
After obtaining approval from Ethical Review Committee (ERC) of Aga Khan University Hospital Karachi (AKUH) and inform about the study to primary surgeon (who ever doing the surgical procedure on this time), informed written consent will be obtained from the parents of patients fulfilling the inclusion criteria schedule for surgical procedures on the day before surgery. Assent will be obtained from older children.

The patients will be assigned to one of the two groups by randomization through sealed opaque envelope technique. The envelopes will be prepared using a computer generated randomization table. Randomization envelopes will be used in consecutive order.

Patients will be allocated to either placebo group, who will not receive intravenous paracetamol, or group who will receive intravenous paracetamol.

All patient will be given general anesthesia as per standard of care. Anaesthesia will be standardized as follow. Anaesthesia will be induced by the inhalational route with application of facemask with 8% sevoflurane in 50% oxygen-nitrous oxide mixture. Airway will be managed by laryngeal mask airway (LMA) of appropriate size as recommended by manufacturer and anesthesia will be subsequently maintained with Minimum alveolar concentration 1-2% sevoflurane in 40% oxygen-nitrous mixture with spontaneous ventilation via LMA. Heart rate (HR), noninvasive blood pressure, core body temperature (oral/nasal probe), end-tidal carbon dioxide (ETCO2) and oxygen saturation by pulse oximetry (SpO2) will be monitored throughout.

After induction of anaesthesia, patients will be turned to lateral position and maximum safe dose of ropivacaine will be calculated (3mg/kg) and documented. After all aseptic measures, butterfly needle (size 23 gauge) will be inserted into the sacral hiatus. A total volume of 1 ml/kg of 0.25% ropivacaine solution will be injected in caudal space. The time of performing block will be noted. The success of caudal analgesia will be assessed by monitoring the parameters like heart rate (HR) and blood pressure (BP) in response to incision. In case of tachycardia (>20% from baseline) and hypertension (>20% from baseline), the concentration of sevoflurane will be adjusted. If tachycardia persists for more than 5 minutes despite increasing the sevoflurane concentration, rescue analgesia in the form of fentanyl 1mcg/kg will be administered.

Study drugs will be prepared and dispatch by Clinical Trial Unit (CTU) pharmacy. Eligible consecutive randomized patients belonging to study group will receive intravenous paracetamol approximately about an hour before the end of surgery with a dose of 15mg/kg over 15 to 20 minutes. While the patients belonging to other group will receive placebo. Time of intravenous paracetamol administration will be noted.

After emergence, the children will be taken to the postanesthesia care unit (PACU) where parents will be called to stay with their child. Time of arrival in the recovery room will be noted.The Mean arterial pressures (MAP), heart rate HR, oxygen saturation by pulse oximetry (SPO2), respiratory rate (RR), sedation, agitation, quality and duration of analgesia will be recorded at 15 and 30 minutes and will be followed by 1, 2, 4, and 6 hours following recovery from anaesthesia.

The analgesic status of the patient will be evaluated by trained Research Assistant in the PACU and in the ward by using Children's Hospital of Eastern Ontario Pain Scale (CHEOPS). This includes crying, facial expression, verbal response, touching the wound and torso and leg movement. It is given in the Appendix.

Sedation will be assessed using a five point scale (0: awake; 1: mild sedation; 2: sleeping, but able to wake; 3: in deep sleep, unable to wake). These observations will be recorded by the same investigator blinded to the medication administered. Same observer will perform the measurements for all patients. A pain score lower than 4 will be considered adequate analgesia. Rescue analgesia will be provided by 0.1 mg/kg i.v. morphine in divided doses (0.025 mg aliquots) and time of doses will be noted on the form.

Analgesia requirement in the postoperative period will be define as a CHEOPS score of 7 or more. Time to the first analgesic requirement will be calculated as the time from the performance of caudal block to the first analgesic dose administered.

Complications like motor block, hypotension and urinary retention will be monitored and recorded in the postoperative period. Modified Bromage Scale will be used to assess motor block i.e 0= No block, 1= Able to move legs, 2= Unable to move legs.

Adverse effects:

Adverse Events are defined as 'Any untoward medical occurrence in a trial patient to whom a research treatment or procedure has been administered, including occurrences which are not necessarily caused by or related to that treatment or procedure.

Adverse effects associated with the paracetamol are rare <1/10000, which includes malaise, increased level of hepatic transaminases and hypersensitivity reaction.

The following data will be collected by an observer in postoperative period: age, weight, height, surgical time, anesthesia time, recovery time, discharge time, need to increase sevoflurane concentration after incision, the need for rescue analgesia in operating room (OR) and PACU, time of voiding urine and time of taking oral fluids, while subjective complaint of heaviness in legs will be asked from children above 3 years only.

SAMPLE SELECTION Inclusion criteria

1. Age 3-10 years
2. American Society of Anesthesiologist class I and II
3. Undergoing hypospadias repair surgery

Exclusion criteria

1. Coagulopathy
2. Aspirin or any other analgesic ingestion in the preceding week
3. Preexisting neurological or spinal disease
4. Hepatic, renal disease and malnutrition

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-10 years
2. ASA (American Society of Anesthesiologists) I and II
3. Undergoing hypospadias repair surgery

Exclusion Criteria:

1. Coagulopathy
2. Aspirin or any other analgesic ingestion in the preceding week
3. Preexisting neurological or spinal disease
4. Hepatic, renal disease and malnutrition
5. Severe hypovolemia
6. Uncontrolled convulsions
7. Refusal of the parents
8. Local Skin infection at the puncture site
9. Allergy to local anesthetics
10. Patient previously involved in other studies

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad S Yousuf, FCPS, Principal Investigator — Aga Khan University
Locations (1):
- Aga Khan University Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hosseini Jahromi SA, Sadeghi Poor S, Hosseini Valami SM, Javadi A. Effects of suppository acetaminophen, bupivacaine wound infiltration, and caudal block with bupivacaine on postoperative pain in pediatric inguinal herniorrhaphy. Anesth Pain Med. 2012 Spring;1(4):243-7. doi: 10.5812/aapm.3551. Epub 2012 Apr 1. PMID 24904808
- [Background] Samuel M, Hampson-Evans D, Cunnington P. Prospective to a randomized double-blind controlled trial to assess efficacy of double caudal analgesia in hypospadias repair. J Pediatr Surg. 2002 Feb;37(2):168-74. doi: 10.1053/jpsu.2002.30247. PMID 11819193
- [Background] Mercan A, Sayin MM, Saydam S, Ozmert S, Tiryaki T. When to add supplemental rectal paracetamol for postoperative analgesia with caudal bupivacaine in children? A prospective, double-blind, randomized study. Paediatr Anaesth. 2007 Jun;17(6):547-51. doi: 10.1111/j.1460-9592.2006.02141.x. PMID 17498016
- [Background] Ozyuvaci E, Altan A, Yucel M, Yenmez K. Evaluation of adding preoperative or postoperative rectal paracetamol to caudal bupivacaine for postoperative analgesia in children. Paediatr Anaesth. 2004 Aug;14(8):661-5. doi: 10.1111/j.1460-9592.2004.01255.x. PMID 15283825
- [Background] Ozbek H, Bilen A, Ozcengiz D, Gunes Y, Ozalevli M, Akman H. The comparison of caudal ketamine, alfentanil and ketamine plus alfentanil administration for postoperative analgesia in children. Paediatr Anaesth. 2002 Sep;12(7):610-6. doi: 10.1046/j.1460-9592.2002.00913.x. PMID 12358657
- [Background] Gunter JB. Benefit and risks of local anesthetics in infants and children. Paediatr Drugs. 2002;4(10):649-72. doi: 10.2165/00128072-200204100-00003. PMID 12269841
- [Background] Mohammed BS, Engelhardt T, Cameron GA, Cameron L, Hawksworth GM, Hawwa AF, McElnay J, Helms PJ, McLay JS. Population pharmacokinetics of single-dose intravenous paracetamol in children. Br J Anaesth. 2012 May;108(5):823-9. doi: 10.1093/bja/aes025. Epub 2012 Mar 1. PMID 22389380
- [Background] Perrott DA, Piira T, Goodenough B, Champion GD. Efficacy and safety of acetaminophen vs ibuprofen for treating children's pain or fever: a meta-analysis. Arch Pediatr Adolesc Med. 2004 Jun;158(6):521-6. doi: 10.1001/archpedi.158.6.521. PMID 15184213
- [Background] Prins SA, Van Dijk M, Van Leeuwen P, Searle S, Anderson BJ, Tibboel D, Mathot RA. Pharmacokinetics and analgesic effects of intravenous propacetamol vs rectal paracetamol in children after major craniofacial surgery. Paediatr Anaesth. 2008 Jul;18(7):582-92. doi: 10.1111/j.1460-9592.2008.02619.x. Epub 2008 May 8. PMID 18482233
- [Background] Nnaji CT, Onajin-Obembe B, Ebirim L. The analgesic effects of rectal diclofenac versus rectal paracetamol following caudal-bupivacaine for pediatric day-case inguinal herniotomies: a randomized controlled prospective trial. J Pediatr Surg. 2017 Sep;52(9):1384-1388. doi: 10.1016/j.jpedsurg.2017.05.001. Epub 2017 May 5. PMID 28535959

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Excluded patients n = 5 Parenteral refusal 2, overweight 2, case cancellation 1
Groups:
- Intravenous Paracetamol With Caudal Ropivacaine (Group P): Patients in Group P received Caudal analgesia after the induction of anesthesia, whereas intravenous paracetamol was given approximately an hour before the end of surgery in a dose of 15mg.kg-1 over 15 to 20 minutes
- Placebo (Group C): Normal Saline (0.9%)
Period: Overall Study
Arm/Group | Intravenous Paracetamol With Caudal Ropivacaine (Group P) | Placebo (Group C)
Started | 30 | 29
Completed | 30 | 29
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intravenous Paracetamol With Caudal Ropivacaine: Paracetamol is widely accepted and most commonly used as an adjuvant for postoperative analgesia. It also improves the quality of recovery by attenuating the pain associated with the surgical position. Adverse effects associated with the paracetamol are rare <1/10000, which includes malaise, increased level of hepatic transaminases and hypersensitivity reaction. It has been studied in combination with caudal analgesia with bupivacaine through the rectal route 7,8 with variable results.
  Caudal anaesthesia is effective in alleviating pain below the umbilicus. Also if the caudal block is administered at the beginning of surgery, the effect will start wearing off 2 to 3 hours post surgery. Administration of paracetamol towards end of surgery may help with both these issues. In this study we aim to investigate the effect of adding intravenous paracetamol in combination with caudal analgesia with ropivacaine, hoping that it may improve quality of postoperative analgesia and recovery.
  Paracetamol +caudal ropivacaine: Paracetamol + Ropivacaine
- Total: Total of all reporting groups
Arm/Group | Intravenous Paracetamol With Caudal Ropivacaine | Placebo | Total
Number analyzed (Participants) | 30 | 29 | 59
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5.00 [3.13 to 6.00] | 4.10 [3.11 to 6.00] | 4.60 [3.11 to 6.00]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 30 | 29 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 14.1 [12.1 to 16.3] | 14.8 [14.0 to 16.5] | 14.7 [13.5 to 16.5]
Heart rate [Mean (Standard Deviation); unit: beats per minute] | 104 (13.3) | 103 (16.1) | 103 (14.6)
Surgical Time [Median (Inter-Quartile Range); unit: Minutes] | 65.0 [42.0 to 79.0] | 65.0 [44.3 to 93.0] | 65.0 [42.0 to 90.0]
Anaesthesia Time [Median (Inter-Quartile Range); unit: Minutes] | 109 [76.3 to 128] | 120 [98.0 to 150] | 111 [81.0 to 140]
Blood Pressure (systolic) [Median (Inter-Quartile Range); unit: mmHg] | 99.0 [88.5 to 107] | 92.0 [85.0 to 100] | 95.0 [86.5 to 103]
Blood Pressure (diastolic) [Median (Inter-Quartile Range); unit: mmHg] | 60.0 [45.3 to 63.3] | 51.0 [43.0 to 60.0] | 53.0 [44.0 to 62.0]

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Analgesia Requirement
Description: The requirement of postoperative analgesia of the patient will be evaluated by using Children's Hospital of Eastern Ontario Pain Scale (CHEOPS). This scale has 5 domains. It includes crying, facial expression, verbal response, touching the wound and torso and leg movement. It is a behavioural scale and measures each domain on a numerical scale of 0 to 2. Minimum score is 0 while maximum score is 10. Aggregate score will be added. Score less than 4 will be consider adequate analgesia while score greater than 4 will be consider inadequate analgesia. CHEOPS Pain Score less than four in participants of C and P groups will be reported at different time points.
Time Frame: follow till 6 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Paracetamol With Caudal Ropivacaine (Group P) | Placebo (Group C)
Number analyzed (Participants) | 30 | 29
Participants
  15 minutes | 23 | 25
  30 minutes | 24 | 21
  1 hour | 26 | 25
  2 hour | 30 | 28
  4 hour | 29 | 29
  6 hour | 29 | 29

2. Secondary Outcome: Sedation
Description: Sedation will be assessed by using Pasero Opioid-Induced Sedation Scale (POSS). This scale measures sedation on numerical score of 0 to 4. Minimum score is 0 while maximum score is 4.
  It comprises of; 0: awake; 1: mild sedation; 2: sleeping, but able to wake; 3: Frequently drowsy, arousable, drifts off to sleep during conversation, unable to wake and 4: Somnolent, minimal or no response to verbal or physical stimulation.
  A POSS score of 0, 1, or 2 indicates an acceptable level of sedation, whereas a score of 3 or 4 indicates over-sedation and the need for a reversal agent. This score is just a numerical number with no other value attached to it.
Time Frame: follow till 4 hours postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Paracetamol With Caudal Ropivacaine (Group P) | Placebo (Group C)
Number analyzed (Participants) | 30 | 29
Participants
  Baseline (0-2) | 23 | 23
  Baseline (3-4) | 7 | 6
  30 min (0-2) | 26 | 25
  30 min (3-4) | 4 | 4
  1 hr (0-2) | 30 | 29
  1 hr (3-4) | 0 | 0
  2 hr (0-2) | 30 | 29
  2 hr (3-4) | 0 | 0
  4 hr (0-2) | 30 | 29
  4 hr 3-4 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 6 hours postoperatively.
Arm/Group | Intravenous Paracetamol With Caudal Ropivacaine (Group P) | Placebo (Group C)
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/29
Other Adverse Events (participants affected / at risk) | 0/30 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT03781505/Prot_SAP_000.pdf